CLINICAL TRIAL: NCT00654784
Title: A Phase IIa Double Blind, Randomised, Placebo Controlled, Single Centre Study at the University of Leuven to Assess the Efficacy and Tolerability of Idebenone in 8 - 16 Year Old Males With Cardiac Dysfunction Associated With Duchenne Muscular Dystrophy
Brief Title: Efficacy and Tolerability of Idebenone in Boys With Cardiac Dysfunction Associated With Duchenne Muscular Dystrophy
Acronym: DELPHI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santhera Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNT-II-001
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Results first posted 2011-07-29 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2011-07

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: Duchenne Muscular Dystrophy; DMD; Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — idebenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: idebenone
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: idebenone — idebenone 450 mg/day (150 mg three times a day)
  Arms: 1
Drug: placebo
  Arms: 2

SUMMARY:
Idebenone is a synthetic analogue of coenzyme Q10 and is a powerful antioxidant and essential constituent of the process of energy production on the cellular level. It can protect mitochondria from oxidative damage and boost their impaired function. It is thought that this mechanism will slow decline in heart function that is part of the disease process of Duchenne Muscular Dystrophy (DMD). It is possible that patients may benefit in terms of muscle strength and respiratory function. This pilot trial is designed to investigate this.

ELIGIBILITY:
Inclusion Criteria:

* Patients 8 - 16 years of age at time of enrolment
* Male
* Presence of cardiac involvement/dysfunction, defined by abnormal peak systolic strain in left ventricle (LV) inferolateral wall
* Confirmed diagnosis of DMD (out of frame dystrophin gene deletion OR absent/<5% dystrophin protein on muscle biopsy; clinical picture consistent of typical DMD)
* If on chronic glucocorticosteroids treatment (deflazacort, prednisone) for DMD (or any other disease) (i.e. concomitant medication): dosage must be stable (unchanged) 6 months prior to inclusion
* If on chronic medication for DMD associated cardiomyopathy (β-blocker, diuretics): dosage must be stable (unchanged) 3 months prior to inclusion
* Ability to provide reproducible repeat quantitative muscle testing (QMT) upper limb score within 15% of first assessment score (at Visit1/Day 1 versus Screening Visit

Exclusion Criteria:

* Symptomatic cardiomyopathy or heart failure
* Asymptomatic but severe cardiac dysfunction on baseline (Screening) evaluation: Fractional shortening (FS) < 20% and/or Ejection fraction (EF) < 40%
* Use of ACE-inhibitors
* Previous history of ventricular arrhythmias (other than isolated ventricular extrasystole); ventricular arrhythmias presented at Screening
* Previous (6 months or less) participation in any other therapeutic trial for DMD
* Use of coenzymeQ10, idebenone, creatine, glutamine, oxatomide, or any herbal medicines within the last 6 months
* History of significant concomitant illness or significant impairment of renal or hepatic function
* Known individual hypersensitivity to idebenone

Ages: 8 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2005-10; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Buyse, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Children's Hospital, University Hospital, Leuven, Belgium

REFERENCES:
- [Result] Buyse GM, Goemans N, van den Hauwe M, Thijs D, de Groot IJ, Schara U, Ceulemans B, Meier T, Mertens L. Idebenone as a novel, therapeutic approach for Duchenne muscular dystrophy: results from a 12 month, double-blind, randomized placebo-controlled trial. Neuromuscul Disord. 2011 Jun;21(6):396-405. doi: 10.1016/j.nmd.2011.02.016. Epub 2011 Mar 23. PMID 21435876

RESULTS

PARTICIPANT FLOW:
Groups:
- Idebenone 450 mg/ Day: idebenone 150 mg tablet: One tablet 3 times a day (Tid) with meals
- Placebo: Placebo tablet: One tablet 3 times a day (Tid) with meals
Period: Overall Study
Arm/Group | Idebenone 450 mg/ Day | Placebo
Started | 13 | 8
Completed | 13 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Idebenone 450 mg/ Day | Placebo | Total
Number analyzed (Participants) | 13 | 8 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 8 | 21
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 13.4 (2.1) | 10.8 (1.9) | 12.4 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 8 | 21
Region of Enrollment [Number; unit: participants]
  Belgium | 13 | 8 | 21

OUTCOME MEASURES:

1. Primary Outcome: The Relative Change in Peak Systolic Radial Strain of the Left Ventricle (LV) Inferolateral Wall From Baseline (at Screening) to Week 52, Assessed by Color Doppler Myocardial Imaging (CDMI).
Description: * Assessing the peak systolic radial strain of the left ventricle inferolateral wall is used to characterize the cardiac involvement in the DMD patients.
  * Color Doppler Myocardial Imaging technique is used to quantify regional myocardial function.
  The cardiac involvement in DMD is characterized by degeneration, atrophy and fibrosis of the myocardium, leading to dilated cardiomyopathy. The process begins in the posterolateral wall of the left ventricle, with septal involvement appearing at later stages.
Time Frame: baseline and Week 52
Population: At Week 52, data from only 18 patients were available for the primary endpoint analysis due to missing data from 2 patients and the inability to acquire data from a 3rd patient. The efficacy comparison for the primary endpoint was conducted using the LOCF method in the ITT population. In addition, the analysis was repeated using the OC dataset.
Measure: Mean (Standard Deviation); unit: % change in peak systolic
Arm/Group | Idebenone 450 mg/ Day | Placebo
Number analyzed (Participants) | 11 | 7
% change in peak systolic | 104.4 (92.0) | 28.9 (40.7)

2. Secondary Outcome: Respiratory Function: Forced Vital Capacity (FVC), Forced Expiratory Volume in 1 Second (FEV1), Maximal Inspiratory Pressure (MIP) and Peak Flow (PF)
Time Frame: 1 year
Reporting Status: Not Posted

3. Secondary Outcome: Skeletal Muscle Strength (Upper Limb, Right and Left): Hand Grip, Elbow Flexors and Elbow Extensors (Upper Limb Score) Timed Walking Test (10 Metres) (Ambulant Patients Only)
Time Frame: 1 year
Reporting Status: Not Posted

4. Secondary Outcome: Safety and Tolerability, Assessed by Adverse Events, Blood and Urine Laboratory Measures, ECG.
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Idebenone 450 mg/ Day | Placebo
Serious Adverse Events (participants affected / at risk) | 1/13 | 1/8
Other Adverse Events (participants affected / at risk) | 12/13 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idebenone 450 mg/ Day (N=13) | Placebo (N=8)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idebenone 450 mg/ Day (N=13) | Placebo (N=8)
Gastrointestinal disorders (Gastrointestinal disorders) | 4 (5) | 5 (6)
Infections (Infections and infestations) | 8 (19) | 5 (12)
General disorders (General disorders) | 2 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No